CLINICAL TRIAL: NCT03322397
Title: Study of Daily Life and Health
Brief Title: Adolescent Acts of Kindness Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Andrew J. Fuligni, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 17-001018
Record Dates: First submitted 2017-10-23; First posted 2017-10-26 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Inflammation; Mental Health Wellness 1
Keywords: adolescence; immune function; gene expression; psychological well-being; social connection; kindness
MeSH Terms: conditions — Inflammation; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: 90 participants will randomly be assigned to one of three interventions. Participants will complete a 4-week intervention. All outcomes will be measured before and after the intervention, and some psychological measures will be collected weekly throughout the intervention.
Who Masked: Participant
Masking Description: Participants will be told that the investigatos are studying the daily lives of teens. They will not be informed of the other arms of the experiment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kindness to Others (Experimental): Participants will complete the 'Other-Focused Acts of Kindness Intervention' by performing acts of kindness for others. They be asked to complete 3 kind acts for others throughout the week for 4 weeks. They will receive text messages three days per week (either Tuesday, Thursday, and Saturday or Wednesday, Friday, and Sunday) and will report on their kind act later that day.
  Interventions: Behavioral: Other-Focused Acts of Kindness Intervention
- Kindness to Self (Active Comparator): Participants will complete the 'Self-Focused Acts of Kindness Intervention' by performing acts of kindness for themselves. They be asked to complete 3 kind acts for others throughout the week for 4 weeks. They will receive text messages three days per week (either Tuesday, Thursday, and Saturday or Wednesday, Friday, and Sunday) and will report on their kind act later that day.
  Interventions: Behavioral: Self-Focused Acts of Kindness Intervention
- Daily Report (Sham Comparator): Participants will complete the 'Daily Reports' and be asked to report their daily activities throughout the week for 4 weeks. They will receive text messages three days per week (either Tuesday, Thursday, and Saturday or Wednesday, Friday, and Sunday) and will list activities from their day.
  Interventions: Behavioral: Daily Reports

INTERVENTIONS:
Behavioral: Self-Focused Acts of Kindness Intervention — Participants engage in positive behaviors by completing acts of kindness for themselves three times per week. These acts should require effort and be outside of an individual's normal routine.
  Arms: Kindness to Self
Behavioral: Other-Focused Acts of Kindness Intervention — Participants engage in positive behaviors by completing acts of kindness for others three times per week. These acts should require effort and be outside of an individual's normal routine.
  Arms: Kindness to Others
Behavioral: Daily Reports — Participants will report their daily activities three times per week. Aside from reporting at the end of the day, no changes should be made to the individual's normal routine.
  Arms: Daily Report

SUMMARY:
Adolescents will complete a 4-week intervention, during which they will either complete a kind act for others, complete a kind act for themselves, or report their daily activities three days per week. Psychological and physiological measures will be indexed before and after the intervention.

DETAILED DESCRIPTION:
Stress and early adversity have been found to influence immune function via enhanced expression of the conserved transcriptional response to adversity (CTRA) genetic profile. Expression of this genetic profile was reduced in adults who completed a prosocial behavior intervention. This project aims to implement this intervention in adolescents. 90 high school students will be recruited and assigned to one of three groups (30/group). Participants will either conduct 3 acts of kindness for themselves, conduct 3 acts of kindness for others, or report about their day 3 times per week for 4 weeks. During this intervention, they will receive text messages 3 days per week instructing them to complete their respective act. Participants will provide a brief description of this act that evening, as well as complete brief surveys at the end of the week for each week of the intervention. Participants will come into the lab twice, once before and once after the 4-week intervention. During these lab sessions participants will complete survey measures, have their heart rate measured, and have a blood draw conducted by a trained phlebotomist. Participants' parents will also complete a brief survey to provide demographic information and an idea of what prosocial behaviors participants witnessed in their home. The investigators will use these data to assess the effects of prosocial behavior on health and the psychological mechanisms underlying these effects. At the second study visit, participants will be given the opportunity to donate part of their study payment to a charity to measure prosociality. Any donations will be vetted with the psychology department's accounting group prior to making any donations in the university's name. Scott Monatlik, Director, Tax and Information Practices, at smonatlik@finance.ucla.edu or (310) 794-6724 will be contacted and information regarding the appropriate steps to take to ensure that the donation is made to an acceptable charity prior to any donations. Actual helping behavior (donations) is measured to provide an ecologically valid experimental evaluation of prosociality rather than traditional metrics of computerized, fictional giving. Conceptual frameworks from developmental and health psychology guide the hypothesis that prosocial behavior will influence adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 14-17

Exclusion Criteria:

* None

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2017-10-08 (Actual); Primary Completion 2019-01-13 (Actual); Study Completion 2019-01-13 (Actual)

PRIMARY OUTCOMES:
Average Positive Affect | Weekly over 5 weeks
  Average Positive Affect as assessed by the positive affect subscale of the Affect Adjective Checklist. An average is taken across four items, and scores range from 1 to 5 with higher scores indicating more positive affect over the week.

SECONDARY OUTCOMES:
Inflammatory Gene Expression | Baseline and one-week post intervention (elapsed time of 5 weeks)
  Change in inflammatory gene expression from baseline to one week following the intervention as assessed by assays of the conserved transcriptional response to adversity profile of gene expression in leukocytes.
Average Psychological Flourishing | Baseline and one-week post intervention (elapsed time of 5 weeks)
  Change in average psychological flourishing from baseline to one week following the intervention as assessed by Mental Health Continuum-Short Form at week 5. An average is taken across 20 items, and scores range from 1 to 6, with higher values representing greater psychological flourishing.
Average Negative Affect | Weekly over 5 weeks
  Average negative affect as assessed by the negative affect subscale of the Affect Adjective Checklist. An average is taken across five items, and scores range from 1 to 5 with higher scores indicating more negative affect over the week.

OTHER OUTCOMES:
Average Stress | Weekly over 5 weeks
  Average stress as assessed by the Perceived Stress Scale. An average is taken across 10 items, and scores range from 1 to 5 with higher scores indicating greater stress.
Sleep Quality | Weekly over 5 weeks
  Sleep quality as assessed by the Pittsburgh Sleep Quality Index (PSQI). The assessment has 7 components, each scored from 0 to 3. A sum is taken across these components, such that total scores range from 0 to 21 with higher scores indicating poorer sleep.
Inflammatory Composite | Baseline and one-week post intervention (elapsed time of 5 weeks)
  Change in inflammation from baseline to one week following the intervention as assessed by the concentration of a variety of inflammatory cytokines (e.g., IL-6, IL-1).
Respiratory Sinus Arrythmia (RSA) | Baseline and one-week post intervention (elapsed time of 5 weeks)
  Change in RSA from baseline to one week following the intervention as assessed by high-frequency heart rate variability during paced breathing.
Average Social connection | Weekly over 5 weeks
  Average social connection as assessed by the relatedness subscale of the Balanced Measure of Psychological Needs. An average is taken across 6 items, and scores range from 1 to 5 with higher scores indicating greater social connection.
Donation | 5 weeks
  Donation as assessed by the amount of money participants donated (maximum of $10) to a charity for foster youth.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Fuligni, PhD, Principal Investigator — Professor
Locations (1):
- Adolescent Development Lab at UCLA, Los Angeles, California, United States